CLINICAL TRIAL: NCT05449132
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Trial, to Evaluate the Efficacy and Safety of a Single Intra-articular Injection of RTX-GRT7039 in Adult Subjects With Pain Associated With Osteoarthritis of the Knee
Brief Title: Comparison of a Single RTX-GRT7039 and Placebo Intra-articular Injection for Pain Associated With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF7039-02; 2021-005020-38 (EudraCT Number); U1111-1268-7267 (Other: Universal Trial Number)
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
Keywords: Knee; Osteoarthritis; Pain assessment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RTX-GRT7039 (Experimental): Participants will receive a intra-articular injection of RTX-GRT7039 during the 52-week double-blind treatment period.
  Interventions: Drug: RTX-GRT7039
- Placebo (Placebo Comparator): Participants will receive a intra-articular injection of placebo matching RTX-GRT7039 during the 52-week double-blind treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RTX-GRT7039 — RTX-GRT7039 intra-articular injection.
  Arms: RTX-GRT7039
Drug: Placebo — Placebo matching RTX-GRT7039 intra-articular injection.
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, parallel-group, multi-site, clinical trial to confirm the efficacy and safety of single injection of RTX-GRT7039 versus placebo in patients who have pain associated with osteoarthritis of the knee despite standard of care.

DETAILED DESCRIPTION:
This trial comprises a total observation period of up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has given written informed consent to participate.
* The participant is 18 years of age or older at the Screening Visit.
* The participant has a diagnosis of osteoarthritis of the knee based on American College of Rheumatology criteria and functional capacity class of I to III.
* There is a documented history indicating that participant has insufficient pain relief with previous Standard of Care.

Exclusion Criteria:

* The participant has past joint replacement surgery of the index knee.
* The participant has a history of significant trauma or surgery (e.g., open or arthroscopic) to the index knee within 12 months of Screening.
* The participant has periarticular pain from any cause other than osteoarthritis, including referred pain, bursitis, or tendonitis.
* The participant has clinical hip osteoarthritis on the side of the index knee.
* The participant has pre-existing osteonecrosis, subchondral insufficiency fracture, atrophic osteoarthritis, severe bone on bone osteoarthritis, knee pain attributable to disease other than osteoarthritis, or the participant has rapidly progressing osteoarthritis (RPOA) Type I or Type II.
* The participant has significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the target knee (varus >10, valgus >10) by X-ray as assessed by independent Central Readers at Screening Visit.
* The participant has other conditions that could affect trial endpoint assessments of the index knee.
* The participant has current clinically significant disease(s) or condition(s) that may affect efficacy or safety assessments, or any other reason which, in the investigator's opinion, may preclude the participant's participation in the full duration of the trial.
* The participant has a history of hypersensitivity to resiniferatoxin (RTX) or any similar component (capsaicin, chili peppers).
* The participant is currently participating or was participating in another investigational drug trial within 3 months prior to the Screening Visit.
* The participant is an employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site or is a family member of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score | From Baseline up to Week 12
  The WOMAC pain subscale will be assessed using an 11-point numeric rating scale (NRS), where 0= no pain and 10=worst pain imaginable.

SECONDARY OUTCOMES:
Change from Baseline in WOMAC Pain Subscale Score | From Baseline up to Week 52
  The WOMAC pain subscale will be assessed using an 11-point NRS, where 0= no pain and 10=worst pain imaginable.
Change from Baseline in WOMAC Physical Function Subscale Score | From Baseline up to Week 52
  The WOMAC physical function subscale will be assessed using 11-point NRS, where 0= no difficulty and 10=extreme difficulty.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | From Baseline up to Week 52
Change from Baseline in WOMAC Stiffness Subscale Score | From Baseline up to Week 52
  The WOMAC stiffness subscale will be assessed using an 11-point NRS, where 0= no stiffness and 10= extreme stiffness.
Change from Baseline in WOMAC Total Score | From Baseline up to Week 52
  The WOMAC total score will be calculated as the sum of pain subscale score, stiffness subscale score and physical function subscale score. It will be calculated by averaging all of the scores available for the questions and assessed using an 11-point NRS, where 0=better outcome and 10=worst outcome.
Change from Baseline in WOMAC A1 (Walking Pain) Subscale Score | From Baseline up to Week 52
  The WOMAC A1 subscale will be assessed using an 11-point NRS, where 0= no pain and 10=worst pain imaginable.
Percentage of Participants With at Least 30%, 50% and 70% Reduction From Baseline in WOMAC Pain Subscale Score | From Baseline up to Week 52
  The WOMAC pain subscale will be assessed using an 11-point NRS, where 0= no pain and 10=worst pain imaginable.
Percentage of Participants With at Least 30%, 50% and 70% Reduction From Baseline in WOMAC A1 (Walking Pain) Subscale Score | From Baseline up to Week 52
  The WOMAC A1 subscale will be assessed using an 11-point NRS, where 0= no pain and 10=worst pain imaginable.
Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response | From Baseline up to Week 52
  OMERACT-OARSI response: A high improvement of >=50% (percentage change) and >=2 (absolute change) in either the WOMAC pain subscale score or WOMAC physical function subscale score, OR an improvement in at least 2 of the following 3:
  * Improvement of >=20% (percentage change) and >=1 (absolute change) in the WOMAC pain subscale score.
  * Improvement of >=20% (percentage change) and >=1 (absolute change) in the WOMAC physical function subscale score.
  * Improvement of >=20% (percentage change) and >=10 (absolute change) in Patient Global Assessment (PGA) of osteoarthritis. Absolute values will be normalized to the 0 (no pain) to 100 scale (higher pain/difficulty).
Percentage of Participants Categorized by Each Patient Global Impression of Change (PGIC) Score | From Baseline up to Week 52
  The 7-point PGIC is a complementary assessment of analgesic efficacy on a 7-point scale where 1 = "Very much improved" and 7 = "Very much worse".
Change From Baseline in EuroQol-5 Dimension Health Questionnaire 5 Levels (EQ-5D-5L) Score | From Baseline up to Week 52
  EQ-5D consists of EQ-5D descriptive system (Index score) and EQ visual analogue scale (VAS). EQ-5D-5L Index Score ranges from 0 to 1, with 0 representing death and 1.0 representing perfect health. EQ-5D-5L-VAS records participant's self-rated health on a vertical VAS that range from 0 (worst imaginable) to 100 (best imaginable).
Change From Baseline in 36-Item Short-Form (SF-36) Domain Scores | From Baseline up to Week 52
  The SF-36 domain scores range from 0 (worst value) to 100 (best value), with higher scores reflecting better health status.
Number of Participants Reporting Durability of Effect | From Baseline up to Week 52
  Durability of effect is defined as time from an improvement in WOMAC pain subscale to pain recurrence. Pain recurrence is defined as no reduction of >=30% from baseline in the WOMAC Pain subscale score (assessed using an 11-point NRS, where 0= no pain and 10=worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (80):
- United States (55):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Associates (AARA) P.C, Glendale, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Tucson Orthopaedic Research Center, Tucson, Arizona
  - Orange County Research Institute, Anaheim, California
  - Core Health Care Group, Cerritos, California
  - Acclaim Clinical Research, Inc., San Diego, California
  - Dr. Hans Richard Barthel, MD Office Of, Santa Barbara, California
  - Medvin Clinical Research, Thousand Oaks, California
  - Westlake Medical Research, Thousand Oaks, California
  - Allied Biomedical Research Institute, Miami, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Vista Clinical Research, Newnan, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Injury Care Research, Boise, Idaho
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - Chicago Medical Research, LLC, Hazel Crest, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - LCMC Health Urgent Care - Lakeview, New Orleans, Louisiana
  - June DO,PC, Lansing, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Accellacare Research of Charlotte, Charlotte, North Carolina
  - Park Road Medical Clinic, Charlotte, North Carolina
  - Accellacare of Raleigh, Raleigh, North Carolina
  - Raleigh Medical Group, Raleigh, North Carolina
  - Accellacare Research of Winston Salem, Winston-Salem, North Carolina
  - Gastroenterology Associates of the Piedmont, Winston-Salem, North Carolina
  - The Center For Clinical Research, Winston-Salem, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Antria Inc., Indiana, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Chan Soon-Shiong Medical Center at Windber, Windber, Pennsylvania
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Accellacare - Knoxville, Knoxville, Tennessee
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research Center LLC, Charlottesville, Virginia
- Denmark (2):
  - Arthroscopic Center, Copenhagen University Hospital, Amager
  - The Parker Institute-Frederiksberg Hospital, Frederiksberg
- Portugal (3):
  - Hospital de Cascais, Alcabideche
  - Hospital Dos Lusiadas Lisboa, Lisbon
  - Hospital CUF Porto, Porto
- Spain (14):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Sanitas Cima, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitaro De Elche, Elche
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de La Princesa, Madrid
  - Accellacare Alcobendas, Madrid
  - Hospital Universitario Virgen De La Arrixaca (Huva), Murcia
  - Consorci Corporacio Sanitaria Parc Tauli, Sabadell
  - Institut d Investigacio i Innovacio Parc Tauli, Hospital Universitari Parc Tauli, Sabadell
  - Clinica Gaias, Santiago de Compostela
  - Complexo Hospitalario Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Clinico Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Quironsalud Infanta Luisa, Seville
- United Kingdom (6):
  - Accellacare-Northamptonshire, Corby, Northamptonshire
  - Robert Jones & Agnes Hunt Orthopaedic Hospital - Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Powys
  - Royal Orthopaedic Hospital - Nhs Foundation Trust, Birmingham
  - Glasgow Royal Infirmary - Greater Glasgow Health Board, Glasgow
  - Accellacare North London, Northwood
  - Accellacare South London, Orpington

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Data Sharing Principles.
URL: https://www.grunenthal.com/en/research-and-development/clinical-trials/data-sharing-clinical-trials